CLINICAL TRIAL: NCT00841360
Title: A Pilot Study to Identify Undiagnosed Asymptomatic HIV Infections in Adolescent and Young Adult Women
Brief Title: ID and Testing Via Friendship Networks
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 067
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: Asymptomatic HIV; HIV Infections
Keywords: Social network; Asymptomatic HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- HIV Positive: Participant self-discloses as HIV positive.
  Sexually experienced females between the ages of 13 and 24 years old and of African American race, Hispanic/Latina ethnicity, or mixed-race/ethnicity, which must include African American race and/or Hispanic/Latina ethnicity.
  Interventions: Other: Index Recruiter
- HIV Negative: Participant self-discloses as HIV negative (based on receiving a negative HIV test within 12 months prior to study consent).
  Sexually experienced females between the ages of 13 and 24 years old and of African American race, Hispanic/Latina ethnicity, or mixed-race/ethnicity, which must include African American race and/or Hispanic/Latina ethnicity.
  Interventions: Other: Index Recruiter
- HIV Status Unknown: Participant self-discloses as HIV negative (no history of prior HIV testing, or HIV screening more than 12 months prior to date of study consent).
  Sexually experienced females between the ages of 13 and 24 years old and of African American race, Hispanic/Latina ethnicity, or mixed-race/ethnicity, which must include African American race and/or Hispanic/Latina ethnicity.
  Interventions: Other: Index Recruiter
- Friendship Network Members: Friendship network members will also consist of sexually experienced females, aged 13 years and older. Although most members are expected to be of African American race and/or Hispanic/Latina ethnicity, all races and ethnicities will be included.
  Interventions: Other: Friendship Network Member

INTERVENTIONS:
Other: Index Recruiter — Participants agree to recruit at least two female friends from their friendship network to undergo HIV screening.
  Groups: HIV Negative; HIV Positive; HIV Status Unknown
Other: Friendship Network Member — Participants are recruited by Index Recruiters to enroll in study and receive HIV screening and complete a questionnaire either on Facilitators of HIV Screening or Barriers to HIV Screening.
  Groups: Friendship Network Members

SUMMARY:
This is a pilot study with a cross-sectional research design to recruit Hispanic/Latina and African American adolescent and young adult women, aged 13-24 years to serve as index recruiters, who will in turn recruit members of her female friendship network, aged 13 years and older to undergo HIV screening. This approach seeks to identify new HIV infections in the target population.

DETAILED DESCRIPTION:
The proposed pilot study will utilize a cross-sectional research design to recruit Hispanic/Latina and African American young women to undergo HIV screening. The research design will consist of a friendship-based, female network recruitment approach that incorporates a dual method of incentives for index recruiters and network members as a strategy for identifying new HIV infections in the target population. Among sexually experienced young women (many of whom who reside in communities with a high prevalence of STIs and HIV), 50 who self-identify as HIV positive, 50 who self-identify as HIV negative (based on receiving a negative HIV test within 12 months prior to study consent), and 50 whose HIV status is self-reported as unknown (who have no history of prior HIV testing or who had HIV screening more than 12 months prior to date of study consent) will be recruited. These women will serve as index recruiters to recruit two or more (on average four) female friendship network members to undergo HIV screening. The index recruiters will be recruited through three participating ATN sites utilizing the existing infrastructure within the AMTUs and their community and clinical partnerships. Index participants that agree to take part in this research will be asked to self-disclose their HIV status, to complete a risk assessment and indicate their willingness to recruit their close female friends to undergo HIV screening. In addition, index recruiters who self-identify as HIV negative and those who do not know their HIV status will be invited to undergo HIV screening.

Index recruiters will be given up to four months to recruit members of their friendship network. At the end of this recruitment period or after successful recruitment of two or more friendship network members, whichever comes first, all index recruiters will be asked to complete a brief questionnaire that describes factors that both facilitated and hindered their ability to recruit the friendship network members. Sexually experienced friendship network members who agree to participate in the study will also complete a risk assessment regardless of whether or not they agree to undergo HIV screening. Participation in this study will be strictly on a voluntary basis.

ELIGIBILITY:
Inclusion Criteria for INDEX RECRUITERS:

* Born female;
* Aged 13-24 years at the time of consent;
* African American or Hispanic/Latina ethnicity or mixed-race/ethnicity, which must include African American race and/or Hispanic/Latina ethnicity;
* A history of sexual intercourse with at least one male sexual partner;
* Any HIV status as follows: (1) HIV positive; (2) HIV negative defined as receiving a negative HIV test result < 12 months prior to the date of study consent); or (3) HIV status unknown defined as either no history of HIV testing or receipt of negative HIV test results more than 12 months prior to the date of study consent);
* History of vaginal and/or anal sexual intercourse with a male;
* Willing to complete a HIV risk assessment; and
* Willing to recruit two or more friendship network members to discuss and eventually undergo HIV screening;
* Ability to understand written and spoken English; and
* Willing to provide written informed consent/assent.

Inclusion Criteria for FRIENDSHIP NETWORK MEMBERS:

* Born female;
* Aged > 13 years at the time of consent;
* A history of sexual intercourse with at least one male sexual partner;
* Willing to complete an HIV risk assessment;
* Willing to discuss and consider HIV screening;
* Self-report that the most recent HIV test result was negative, or has no prior history of HIV testing;
* Ability to understand written and spoken English; and
* Willing to provide written informed consent/assent.

Exclusion Criteria for INDEX RECRUITERS:

* Psychiatric disorder (untreated) associated with thought disorder, hallucinations, acute substance use withdrawal. Stabilized patients receiving appropriate psychiatric care will not be excluded if informed consent can be reasonably assumed;
* Visibly distraught and/or visibly emotionally unstable (e.g., depressive mood; exhibiting manic, suicidal, or violent behavior);
* Active drug or alcohol use or dependence that, in the opinion of the site personnel, would interfere with ability to give true informed consent and to adhere to the study requirements; and
* Acutely ill at the time of enrollment.

Exclusion Criteria for FRIENDSHIP NETWORK MEMBERS:

* Self-report an HIV positive test result;
* Psychiatric disorder (untreated) associated with thought disorder, hallucinations, acute substance use withdrawal. Stabilized patients receiving appropriate psychiatric care will not be excluded if informed consent can be reasonably assumed;
* Visibly distraught and/or visibly emotionally unstable (e.g., depressive mood; exhibiting manic, suicidal, or violent behavior);
* Active drug or alcohol use or dependence that, in the opinion of the site personnel, would interfere with ability to give true informed consent and to adhere to the study requirements;
* Acutely ill at the time of enrollment.

Ages: 13 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Index recruiters will consist of sexually experienced females between the ages of 13 and 24 years old and of African American race, Hispanic/Latina ethnicity, or mixed-race/ethnicity, which must include African American race and/or Hispanic/Latina ethnicity.
  Friendship network members will also consist of sexually experienced females, aged 13 years and older. Although most members are expected to be of African American race and/or Hispanic/Latina ethnicity, all races and ethnicities will be included.
Sampling Method: Non-Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Number of young women (HIV status positive, negative, or unknown) who are identified and recruited to serve as index recruiters divided by the number of young women screened. | 2
Proportion of index recruiters who recruit two or more of their female, friendship network members to undergo HIV screening. | 2 years
A description of factors that facilitate and hinder index recruiters in recruiting female friendship network members. | 2 years
A description of factors that facilitate and hinder HIV screening among female friendship network members. | 2 years
A preliminary estimate of HIV infection prevalence among the friendship networks of all index recruiters and separately in the friendship networks of each group of index recruiters. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cherrie B Boyer, PhD, Study Chair — University of California, San Francisco; ATN
Locations (3):
- United States (3):
  - University of Miami School of Medicine, Miami, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- See also: ATN Website — https://www.atnonline.org/